CLINICAL TRIAL: NCT06626919
Title: A Phase 1 Study of Anitocabtagene Autoleucel for the Treatment of Subjects With Non-oncology Plasma Cell-related Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arcellx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC-311
Record Dates: First submitted 2024-09-19; First posted 2024-10-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Muscular Diseases; Neuromuscular Manifestations; Autoimmune; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Myasthenia Gravis; Muscle Weakness
Keywords: ARC-311; CART; CAR-T; BCMA; Anito-cel; Generalized Myasthenia Gravis; gMG; MG; Myasthenia Gravis; non-oncology plasma cell; autoimmune; auto-antibody; chimeric antigen receptor; D-Domain chimeric antigen receptor; B-cell maturation antigen (BCMA); anitocabtagene autoleucel
MeSH Terms: conditions — Muscular Diseases; Neuromuscular Manifestations; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Myasthenia Gravis; Muscle Weakness | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- anito-cel (Experimental): Single dose of anito-cel cells infused intravenously
  Interventions: Biological: anito-cel; Drug: Standard Lymphodepletion regimen

INTERVENTIONS:
Biological: anito-cel — Anitocabtagene autoleucel BCMA directed CAR T-cell therapy using a novel, synthetic binding domain, called a D-Domain
  Other Names: anitocabtagene autoleucel; CART-ddBCMA
Drug: Standard Lymphodepletion regimen — Standard lymphodepletion regimen subject receive 5 days prior to CAR T infusion
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
A Phase 1 dose-escalation study designed to evaluate the safety, tolerability, and preliminary efficacy of anito-cel in subjects with generalized myasthenia gravis (GMG). Anitocabtagene autoleucel (anito-cel) is a BCMA-directed CAR-T cell therapy.

DETAILED DESCRIPTION:
This is a Phase 1 open-label, multi-center safety and dose-escalation study of anito-cel* in adult subjects with GMG (MGFA Grade 2 to 4a), in whom immunosuppressive therapy is clinically indicated in the judgement of the treating neurologist. The primary objective of this study is to assess the safety profile, including any DLT and identification of a MTD (if applicable), to support selection of the RP2D of anito-cel when administered to subjects with GMG.

The study will have the following sequential phases: screening, enrollment (leukapheresis), pretreatment with lymphodepletion (LD) chemotherapy, treatment with anito-cel and follow-up. Optional bridging therapy is allowed at investigator discretion while anito-cel is being manufactured.

Following a single infusion of anito-cel both safety and efficacy data will be assessed. The DLTs will be assessed in the first 28 days following anito-cel administration, and safety data will be collected throughout the study.

*Anitocabtagene autoleucel (anito-cel) drug product consists of autologous T cells that have been genetically modified ex vivo to express a D-domain Chimeric Antigen Receptor (CAR), followed by a cluster of differentiation 8 (CD8) hinge and transmembrane region that is fused to the intracellular signaling domains for 4-1BB and CD3ξ, that specifically recognizes B-cell maturation antigen (BCMA). The active substance of anitocabtagene autoleucel is CAR+ CD3+ T cells that have undergone ex vivo T-cell activation, gene transfer by replication-deficient lentiviral vector, and expansion.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older
* Must have MGFA clinical classification Grades 2-4A at time of screening
* Subject must have clinically active disease and requiring ongoing therapy for GMG
* MG-ADL score 6 and QMG score >10 at screening
* GMG specific autoantibodies must be above the reference laboratory ULN

Exclusion Criteria:

* Subject is pregnant or breastfeeding
* Treatment with Anti-CD20 agents, calcineurin inhibitors, FcRN inhibitors, azathioprine, mycophenolate mofetil, methotrexate, or cyclophosphamide within the specified time frame prior to leukapheresis or prior to anito-cel infusion
* Previous treatment with any gene therapy, chimeric antigen receptor therapy or T cell engager
* Previous thymectomy within 6 months of screening
* Major chronic illness that is not well managed at the time of study entry and in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Assess safety profile, including any DLT and MTD (if applicable) | 24 months
  Type, incidence, and severity of treatment-emergent adverse events (TEAEs), including DLT(s) and laboratory abnormalities
Selection of RP2D | 24 months
  Evaluate the MTD and establish the RP2D

SECONDARY OUTCOMES:
Quantify Clinical Effect of Anito-cel in the Myasthenia Gravis Activities of Daily Living (MG ADL) score | 24 months
  The proportion of subjects achieving a ≥2-point change in the MG ADL score from Baseline at any timepoint after treatment. The MG-ADL is an 8-item patient-reported outcome measure assessing GMG symptoms and functional activities related to activities of daily living and producing a total score ranging from 0 to 24, where higher scores indicate greater severity of disease symptoms.
Quantify Clinical Effect of Anito-cel in the Quantitative Myasthenia Gravis (QMG) score | 24 months
  The proportion of subjects achieving a ≥3-point change in the QMG from Baseline at any timepoint after treatment. The QMG score is a 13-item direct physician assessment scoring system that quantifies disease severity, based on impairments of body functions and structures. The total QMG score ranges from 0 to 39, where higher scores indicate greater disease severity.
Quantify Clinical Effect of Anito-cel in the Myasthenia Gravis Composite (MGC) scale. | 24 months
  The proportion of subjects achieving a ≥3-point change in the MGC score from Baseline at any timepoint after treatment. The MGC is a 10-item assessment that measures signs and symptoms of GMG based on physical examination findings and patient history. The total score ranges from 0 to 50, where higher scores indicate more severe impairment.
Mean change in QMG score | 24 months
  The mean change in the QMG score from Baseline at any timepoint after treatment. The QMG score is a 13-item direct physician assessment scoring system that quantifies disease severity, based on impairments of body functions and structures. The total QMG score ranges from 0 to 39, where higher scores indicate greater disease severity.
Mean change in MG-ADL score | 24 months
  The mean change in the MG-ADLscore from Baseline at any timepoint after treatment. The MG-ADL is an 8-item patient-reported outcome measure assessing GMG symptoms and functional activities related to activities of daily living and producing a total score ranging from 0 to 24, where higher scores indicate greater severity of disease symptoms.
Mean change in MCG score | 24 months
  The mean change in the MGC score from Baseline at any timepoint after treatment. The MGC is a 10-item assessment that measures signs and symptoms of GMG based on physical examination findings and patient history. The total score ranges from 0 to 50, where higher scores indicate more severe impairment.
Mean change in MG-QoL15R score | 24 months
  The mean change in the MG QoL15R score from Baseline at any timepoint after treatment. The MG-QoL15 is a 15-item questionnaire that allows clinicians to estimate a patient's quality of life relevant to GMG. The cumulative scores range from 0 to 60, with higher scores representing decreased quality of life.
Change in titer of myasthenia specific autoantibodies | 24 months
  The proportion of subjects achieving ≥50% reduction in myasthenia-specific autoantibody titers from Baseline at any timepoint after treatment
PK Parameter for anito-cel: Cmax | Day 1 up to 24 months
  Cmax is defined as the maximum observed concentration of anitocel measured/quantified using vector copy number (VCN) on peripheral blood mononuclear cells
PK Parameter for anito-cel: Tmax | Day 1 up to 24 months
  Tmax is defined as the time (observed time point) of Cmax of anitocel measured/quantified using vector copy number (VCN) on peripheral blood mononuclear cells
PK Parameter for anito-cel: Area under the curve (AUC) | Day 1 up to 24 months
  AUC is a measure of the anitocel concentration in the blood measured/quantified using VCN on peripheral blood mononuclear cells over time.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UCLA Medical Center, Los Angeles, California
  - University of California, Irvine, Orange, California
  - Stanford Hospital, Palo Alto, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Columbia University Irving Medical Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas